CLINICAL TRIAL: NCT07302633
Title: Virtual Microscopy Versus Optical Microscopy: Comparison of Two Teaching Methodologies for Achieving Specific Learning Outcomes in Medical Students.
Brief Title: Virtual Microscopy Versus Optical Microscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DR-SADAF-QAMC
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Learning Problem
MeSH Terms: interventions — Microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Students were exposed to optical microscopy (OM); OM is the conventional method of using physical microscopes to examine microscope slides.
  Interventions: Other: Optical Microscopy
- Group II (Experimental): Students were exposed to virtual microscopy (VM); VM is a digital technology that allows students to view and analyze microscope slides through digital platforms.
  Interventions: Other: Virtual Microscopy

INTERVENTIONS:
Other: Optical Microscopy — Students were exposed to optical microscopy (OM); OM is the conventional method of using physical microscopes to examine microscope slides.
  Arms: Group I
Other: Virtual Microscopy — Students were exposed to virtual microscopy (VM); VM is a digital technology that allows students to view and analyze microscope slides through digital platforms.
  Arms: Group II

SUMMARY:
The literature reveals ongoing debate regarding the relative effectiveness of Virtual Microscopy (VM) versus Optical Microscopy (OM) in achieving specific learning outcomes (SLOs). There remains a paucity of comprehensive, comparative research evaluating these methodologies against standardized learning outcomes in the medical undergraduate population. This instigated a comparison of VM and OM as teaching methodologies for pathology in medical education, specifically focusing on their effectiveness in achieving predetermined learning outcomes.

DETAILED DESCRIPTION:
It is now essential to thoroughly evaluate the pedagogical effects of these changing modalities due to the growing trend towards digital learning environments, which has been brought to light by recent global challenges to traditional classroom teaching. By methodically contrasting virtual and optical microscopy for teaching pathology to undergraduate medical students, this work can close this gap. It is anticipated that understanding the superior modality-more especially, how well it achieves predefined learning outcomes-will improve the optimization of pathology instruction in modern medical education and guide evidence-based curriculum selections.

ELIGIBILITY:
Inclusion Criteria:

* Students of either gender
* Aged 20-24 years
* Studying in fourth-year MBBS
* Willing to participate

Exclusion Criteria:

* Students, absent during the interventions or assessments
* Declined or withdrew consent at any stage

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Perceptions and satisfaction | 3 hours
  A five-point Likert scale assessed perceptions and satisfaction with the respective teaching methodology. The likert scale responses were graded as 1 for strongly disagree, 2 for disagree, 3 as neutral, 4 agree, and 5 strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Sadaf Shafique, FCPS, Principal Investigator — Quaid-E-Azam Medical College, Bahawalpur, Pakistan
Locations (1):
- Quaid-E-Azam Medical College, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.